CLINICAL TRIAL: NCT05377905
Title: Phase Ib/II Study of Micro-needle Array Containing Doxorubicin in Immune Competent or Immune-suppressed Patients With Cutaneous Squamous Cell Carcinoma
Brief Title: Microneedle Array Plus Doxorubicin in Cutaneous Squamous Cell Cancer (cSCC)
Acronym: cSCC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Falo, Louis, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Oleg E. Akilov, MD, PhD, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY21090123; 1P50CA254865-01A1 (NIH)
Record Dates: First submitted 2022-05-03; First posted 2022-05-17 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Cutaneous Squamous Cell Carcinoma; Skin Cancers - Squamous Cell Carcinoma
Keywords: micro-needle array; doxorubicin; patch
MeSH Terms: interventions — Doxorubicin; Transdermal Patch

STUDY DESIGN:
Intervention Model Description: This is an open-label, comparative 2-cohort design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Microneedle Array Doxorubicin (MNA-D) (Experimental): Immunocompetent and immuno-incompetent subjects will receive the MNA-D patch on 4 subsequent visits for a 20 minute time period at each application and will include patients who have competent immune systems with cSCC meeting all other inclusion/exclusion criteria and patients considered immuno-incompetent post transplant with cSCC meeting all other inclusion/exclusion criteria.
  Interventions: Drug: Microneedle Array Doxorubicin (MNA-D)

INTERVENTIONS:
Drug: Microneedle Array Doxorubicin (MNA-D) — The Microneedle array patch is loaded/prepared with a total dose of 50 micrograms of Doxorubicin and is applied to a single selected cSCC remnant for a period of 20 minutes for a total of 4 weekly applications
  Other Names: MNA-D; Doxorubicin; Patch

SUMMARY:
The purpose of this study is to test a new method of experimental treatment for cutaneous squamous cell skin cancer, using small adhesive-like patches (a micro-needle applicator or MNA for short), which have dozens of very small micro-needles loaded with extremely low doses of doxorubicin, a chemotherapy agent. The overall goal of this study is to test the safety and effectiveness of these patches. The investigators have established the highest tolerated dose at 50 micrograms in a previous study for a different type of cancer that affects the skin. The investigators will thoroughly evaluate the skin where the patches are applied.

DETAILED DESCRIPTION:
This study will evaluate a novel approach to the treatment of cutaneous squamous cell cancer (cSCC) of patients diagnosed previously by skin biopsy with cSCC utilizing a dissolvable microneedle array (MNA) delivery device that is used to directly and specifically deliver a drug to the tumor microenvironment for skin cancer therapy. The investigators will utilize MNAs to deliver a well-characterized, potent chemotherapeutic agent (doxorubicin) to kill topically accessible, cutaneous SCC cells. In addition to directly killing cancer cells, doxorubicin is known to induce an immunologic cell death with the potential to simultaneously convert a cutaneous neoplasm into a highly potent patient specific immunogen capable of inducing innate, adaptive, and tumor specific effector and memory immune responses. Importantly, doxorubicin is currently in clinical use with a well-established safety profile. It is anticipated that use of the MNA-Doxorubicin (MNA-D) delivery system will enable direct and specific delivery of chemotherapy to the tumor, thereby avoiding any potential for systemic toxicity. The study will be conducted using two groups: one group will consist of patients with immunocompetent immune systems and the second group will consist of patients who have had an organ transplant and are considered immunoincompetent.efficacy and safety evaluation. The first phase is now completed. Following a screening/baseline phase, the MNA-D patch application and assessment visits will occur from week 0 through week 3, followed by a rest week and at week 5, up to week 8, a final follow up visit will take place. At the final follow up visit, the remaining cSCC lesion will be removed in a standard of care manner to ensure that all tissue margins are clear of the cSCC.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a histological diagnosis of cSCC based upon a skin biopsy.
2. Subjects must have resectable stage I-III disease.

   - Measures ≥5 millimeters (mm; post-biopsy) and <100 mm in longest diameter
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2
4. Subjects must have an expected survival of greater than or equal to 12 months.
5. Subjects must not be on any other investigational device/drug treatment.
6. Subjects must be willing to adhere to the instructions of the Investigator and his research team and sign an Informed Consent Form prior to entry into the study.
7. Subjects must have the following pretreatment laboratory parameters: granulocytes ≥1,500/mm3; platelets >50,000/mm3; serum creatinine ≤2X the upper limit of normal (ULN); AST, ALT ≤3X the ULN, bilirubin ≤1.5X ULN unless Gilbert's disease then ≤3X ULN.
8. Subjects must be at least 18 years of age and must be able to understand the written informed consent/assent document.
9. Subjects must have no evidence of active infection, regardless of the degree of severity or localization. Subjects with active infections (whether or not they require antibiotic therapy) may be eligible for study participation after complete resolution of the infection. Subjects on antibiotic therapy must be off antibiotics before beginning treatment.
10. Subjects must not receive any other treatment for cSCC except emollients of subject's choice without topical steroids, anti-fungal or antibacterial topical preparations.
11. Subjects with multiple cSCC may re-enroll in the study if greater than 4 weeks elapses between courses and if all other inclusion/exclusion criteria are met.
12. Patients with HIV infection with CD4+ T-cell (CD4+) counts ≥ 350 cells/uL will be eligible for the study. Patients without a history of AIDS-defining opportunistic infections will be eligible for the study.
13. Subjects must be willing/able to comply with standard of care measures for subjects with cSCC such as sun avoidance and sun protection.

Exclusion Criteria:

1. Subjects with the following tumor characteristics:

   * >4 mm depth;
   * Clark level IV;
   * perineural invasion, lymphovascular invasion;
   * primary site on the ear or non-glabrous lip;
   * location in the hands or feet;
   * large size: ≥10 mm on neck or pretibial area; ≥20 mm on trunk or extremities;
   * indistinct borders;
   * rapid growth;
   * recurrent lesion;
   * lesion in site of chronic inflammation or prior radiation therapy;
   * presence of neurologic symptoms; or • poorly differentiated, and aggressive histopathologic subtypes.
2. Subjects with uncontrolled pain that would preclude participation in the study.
3. Subjects who are pregnant or lactating.
4. Subjects who have sensitivity to drugs that provide local anesthesia.
5. Impaired cardiac function or clinically significant cardiac disease, including any of the following:

   * Symptomatic congestive heart failure requiring treatment
   * Clinically significant cardiac arrhythmia
   * Uncontrolled hypertension
   * Corrected QT interval (QTc) >470 msec at Screening or congenital long QT syndrome
   * Acute myocardial infarction or unstable angina pectoris < 3 months prior to the first dose
   * New York Heart Association Functional Class III or higher (i.e. marked limitation of physical activity due to symptoms, or unable to carry on any physical activity without discomfort)
6. Subjects with other active malignancies with the exception of non-metastatic prostate cancer and carcinoma in situ of the skin and cervix.
7. Active, known, or suspected autoimmune disease or a documented history of autoimmune disease, except vitiligo or resolved childhood asthma/atopy.

   • Individuals with vitiligo, type I diabetes, residual hypothyroidism only requiring hormone replacement, psoriasis not requiring systemic treatment, history of Hashimoto's thyroiditis on stable dose of thyroid hormone replacement therapy, adrenal insufficiency only requiring physiologic steroid replacement, or conditions not expected to recur should not be excluded.
8. Major surgery within 2 weeks of the first dose of study agent
9. History of or current drug-induced interstitial lung disease or pneumonitis Grade ≥2
10. Subjects with the disease only on the face, skin folds, head, scalp, and genital area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events grade 2 or higher to evaluate safety of MNA-D patches in cSCC | Baseline up to week 8
  Evaluated by assessing adverse events grade 2 or higher related to the MNA-D intervention

SECONDARY OUTCOMES:
Change from baseline of local response to the MNA-D patch | Baseline and follow up (weeks 5-8)
  Percentage of tumor clearance of the area directly under the patch is measured..
Tumor clearance from baseline of locoregional (total area of the index lesion) response to the MNA-D Patch | Baseline and follow up (weeks 5-8)
  Percentage of tumor clearance from the entire cSCC lesion treated by the patch is measured including the area directly covered by the MNA and uncovered area of the treated lesion. .
Quantitative pathologic evaluation of tumor depth | Follow up period (weeks 5-8)
  To provide a quantitative assessment of cSCC reduction after treatment, the remnant of cSCC tumors will be excised at week 5-8 and evaluated independently by 2 dermatopathologists in the blinded fashion. The depth of the cSCC will be measured.
Flow cytometry quantitative biologic response evaluation in blood | Baseline and follow up (weeks 5-8)
  Flow cytometry will evaluate in-vivo tumor immune responses in the blood and will analyze total immune activity for increases and/or decreases in T cell populations of interest and other immune cells (e.g., MDSCs, NK cells, B cells, macrophages, dendritic cells) that could influence the frequency and phenotype of these populations.
Flow cytometry quantitative biologic response evaluation in tumor tissue | Baseline and follow up (weeks 5-8)
  Flow cytometry will evaluate in-vivo tumor immune responses in the excised tumor tissue and will analyze total immune infiltrates for increases and/or decreases in T cell populations of interest and other immune cells (e.g., MDSCs, NK cells, B cells, macrophages, dendritic cells) that could influence the frequency and phenotype of these populations.
Percentage of reduction in cSCC tumor | Baseline and follow up (weeks 5-8)
  To provide a quantitative assessment of cSCC reduction after treatment, the remnant of cSCC tumors will be excised at week 5-8 and evaluated independently by 2 dermatopathologists in the blinded fashion. The percentage of reduction in comparison to the original tumor will be reported.
Luminex quantitative biologic response in blood | Baseline and follow up (weeks 5-8)
  Luminex will evaluate in-vivo tumor immune responses for 65 selected serum biomarkers using a multiplex Luminex 100 (Bio-Rad Bio-Plex System) including G-CSF, GM-CSF, IFN-α, IFN-γ, IL-1β, IL-1RA, IL-2, IL-2R, IL-4, IL-5, IL-6, IL- 7, IL-8, IL-10, IL-12, IL-13, IL-15, IL-17, TNF-α, eotaxin, IP-10, MCP-1, MIG, MIP-1α, MIP-1β, RANTES, EGF, FGF-basic, HGF, and VEGF.
Serum SCC-Ag quantitative biologic response in blood | Baseline and follow up (weeks 5-8)
  Serum SCC-Ag levels will evaluate in-vivo tumor immune responses in the blood
Luminex quantitative biologic response evaluation in tumor tissue | Baseline and follow up (weeks 5-8)
  Luminex will evaluate in-vivo tumor tissue immune responses for 65 selected serum biomarkers using a multiplex Luminex 100 (Bio-Rad Bio-Plex System) including G-CSF, GM-CSF, IFN-α, IFN-γ, IL-1β, IL-1RA, IL-2, IL-2R, IL-4, IL-5, IL-6, IL- 7, IL-8, IL-10, IL-12, IL-13, IL-15, IL-17, TNF-α, eotaxin, IP-10, MCP-1, MIG, MIP-1α, MIP-1β, RANTES, EGF, FGF-basic, HGF, and VEGF.
Serum SCC-AG quantitative biologic response evaluation in tumor tissue | Baseline and follow up (weeks 5-8)
  Serum SCC-Ag levels will evaluate in-vivo tumor immune responses in the excised tumor tissue from baseline to week 8

CONTACTS AND LOCATIONS:
Overall Officials: Oleg E Akilov, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madeleine MM, Patel NS, Plasmeijer EI, Engels EA, Bouwes Bavinck JN, Toland AE, Green AC; the Keratinocyte Carcinoma Consortium (KeraCon) Immunosuppression Working Group. Epidemiology of keratinocyte carcinomas after organ transplantation. Br J Dermatol. 2017 Nov;177(5):1208-1216. doi: 10.1111/bjd.15931. Epub 2017 Oct 10. PMID 28994104
- [Background] Hanlon A, Colegio OR. The cutting edge of skin cancer in transplant recipients: scientific retreat of international transplant Skin Cancer Collaborative and Skin Cancer in Organ Transplant Patients Europe. Am J Transplant. 2014 May;14(5):1012-5. doi: 10.1111/ajt.12681. Epub 2014 Mar 10. PMID 24612476
- [Background] Karia PS, Han J, Schmults CD. Cutaneous squamous cell carcinoma: estimated incidence of disease, nodal metastasis, and deaths from disease in the United States, 2012. J Am Acad Dermatol. 2013 Jun;68(6):957-66. doi: 10.1016/j.jaad.2012.11.037. Epub 2013 Feb 1. PMID 23375456
- [Background] Li YY, Hanna GJ, Laga AC, Haddad RI, Lorch JH, Hammerman PS. Genomic analysis of metastatic cutaneous squamous cell carcinoma. Clin Cancer Res. 2015 Mar 15;21(6):1447-56. doi: 10.1158/1078-0432.CCR-14-1773. Epub 2015 Jan 14. PMID 25589618
- [Background] Freeman A, Bridge JA, Maruthayanar P, Overgaard NH, Jung JW, Simpson F, Prow TW, Soyer HP, Frazer IH, Freeman M, Wells JW. Comparative immune phenotypic analysis of cutaneous Squamous Cell Carcinoma and Intraepidermal Carcinoma in immune-competent individuals: proportional representation of CD8+ T-cells but not FoxP3+ Regulatory T-cells is associated with disease stage. PLoS One. 2014 Oct 23;9(10):e110928. doi: 10.1371/journal.pone.0110928. eCollection 2014. PMID 25340823
- [Background] Farasat S, Yu SS, Neel VA, Nehal KS, Lardaro T, Mihm MC, Byrd DR, Balch CM, Califano JA, Chuang AY, Sharfman WH, Shah JP, Nghiem P, Otley CC, Tufaro AP, Johnson TM, Sober AJ, Liegeois NJ. A new American Joint Committee on Cancer staging system for cutaneous squamous cell carcinoma: creation and rationale for inclusion of tumor (T) characteristics. J Am Acad Dermatol. 2011 Jun;64(6):1051-9. doi: 10.1016/j.jaad.2010.08.033. Epub 2011 Jan 20. PMID 21255868
- [Background] Madan V, Lear JT, Szeimies RM. Non-melanoma skin cancer. Lancet. 2010 Feb 20;375(9715):673-85. doi: 10.1016/S0140-6736(09)61196-X. PMID 20171403